CLINICAL TRIAL: NCT00175552
Title: Evaluating the Effectiveness of Different Interpersonal Psychotherapy for Adolescents (IPT-A) Therapist Training Models
Brief Title: Ministry of Child and Family Development (MCFD) Interpersonal Psychotherapy for Adolescents (IPT-A) Training Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: B05-0055; 05-3506
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Education of Therapists Treating Adolescent Depression
Keywords: Depression; Adolescents; IPT; Knowledge translation; Psychotherapy
MeSH Terms: conditions — Depression

INTERVENTIONS:
Behavioral: Psychotherapy Training

SUMMARY:
Evaluating the Effectiveness of Different Interpersonal Psychotherapy for Adolescents (IPT-A) Therapist Training Models

ELIGIBILITY:
Inclusion Criteria:

-adolescent undergoing psychotherapy

Exclusion Criteria:

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Baerg Hall, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia, Canada